CLINICAL TRIAL: NCT04548310
Title: Effect of Muscle Fatigue on Strength, Joint Position Sensation, and Walking in Patients With Multiple Sclerosis
Brief Title: Muscle Fatigue in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Research Assistant, Gazi University
Other Study IDs: 867
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; gait; sensation; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Multiple Sclerosis: MS patients (EDSS: 0-5,5)
  Interventions: Other: Muscles Fatigue
- Healthy group: Healthy individuals without chronic disease
  Interventions: Other: Muscles Fatigue

INTERVENTIONS:
Other: Muscles Fatigue — An exhaustion protocol that reduces knee joint flexor and extensor torque will be applied.

SUMMARY:
It is stated that 85% of patients with Multiple Sclerosis (MS) complain of gait disorders and 35-90% of them have fatigue. Many factors play a role in the fatigue mechanism in MS patients. Fatigue can increase the symptoms that already exist in MS patients. It is thought that fatigue caused a decrease in muscle strength, making walking worse. There are not enough studies investigating whether fatigue affects gait parameters in MS patients.

The aim of this study is to examine the effects of muscle fatigue on muscle strength, joint position sensation, and gait in MS patients.

DETAILED DESCRIPTION:
Patients with MS between 0-5,5 score according to the Extended Disability Status Scale (EDSS) and healthy individuals of similar age and sex to patients will be included in the study. The muscle strength, joint position sensation, gait, and fatigue will be evaluated once.

The investigators will use descriptive statistics and t-tests to compare demographic characteristics between groups and for the categorical variables chi-square. Effect of the group (MS patients or healthy controls), condition (Single task and dual-task conditions), and group × condition interaction will be compared using two-way repeated-measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Participants who 18-65 years of age
* MS patients who are ambulatory (Expanded Disability Status Scale score ≤ 5,5 ) in a stable phase of the disease, without relapses in the last 3 month

Exclusion Criteria:

* Participants who have orthopedic, vision, hearing, or perception problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ambulatory sample
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Knee proprioception | 10 minutes
  Knee proprioception will be evaluated with the active joint reposition test using the isokinetic system (Cybex Norm, Humac, CA, USA).
Knee strength | 20 minutes
  Knee strength will be evaluated using the isokinetic system (Cybex Norm, Humac, CA, USA).
Gait | 5 minutes
  Gait parameters will be assessed via the G-Walk on two separate occasions. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk is built with a triaxial accelerometer 16 bit/axes with multiple sensitivity, a triaxial magnetometer 13 bit and a triaxial gyroscope 16 bit/axes with multiple sensitivity. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.
  Gait symmetry values of the right and left sides are obtained within this report. While the symmetry index ranges from 0 to 100, a value closer to 100 indicates that the gait is more symmetrica.
Perceived Exertion | 1 minute
  The Borg Rating of Perceived Exertion (RPE) scale is a tool for measuring an individual's effort and exertion, breathlessness, and fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Phd, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Suzuki, F. S., Mazuchi, F. A. S., Miranda, M. L. J., Maifrino, L. B. M., Mochizuki, L., & Ervilha, U. F. (2013). What is the most effective protocol to induce fatigue in knee joint muscles? a systematic review. J. Morphol, 30(3), 143-147.